CLINICAL TRIAL: NCT02725476
Title: An Open-label, Single-arm, Pilot Study to Evaluate the Effect of XmAb®5871 on Disease Activity in Patients With IgG4-Related Disease
Brief Title: Study to Evaluate the Effect of XmAb®5871 on Disease Activity in Patients With IgG4-Related Disease (RD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XmAb5871-03
Record Dates: First submitted 2016-03-04; First posted 2016-04-01 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: IgG4-RD
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XmAb5871 (Experimental): XmAb5871 administered by IV infusion for up to a total of 12 infusions
  Interventions: Biological: XmAb5871

INTERVENTIONS:
Biological: XmAb5871

SUMMARY:
The purpose of this Phase 2 study is to investigate the effect of XmAb5871 on IgG4-Related Disease (RD) activity

ELIGIBILITY:
Inclusion Criteria:

* Active IgG4-RD
* Compatible pattern of organ involvement consistent with IgG4-RD that cannot be attributed to other causes
* Histopathologically-proven diagnosis of IgG4-RD
* Peripheral blood plasmablast count >900 cells/mL and/or elevated IgG4-RD levels during screening
* Able and willing to complete the entire study according to the study schedule
* Able and willing to provide written informed consent

Exclusion Criteria:

* History or evidence of a clinically unstable/uncontrolled disorder, condition or disease other than IgG4-RD that, in the opinion of the Investigator would pose a risk to the patient safety or interfere with the study evaluation, procedures or completion
* Malignancy within 5 years (except successfully treated in situ cervical cancer, resected squamous cell or basal cell carcinoma of the skin, or prostate cancer with no recurrence ≥3 years following prostatectomy)
* Presence of recurrent or chronic infections, defined as ≥3 infections requiring antimicrobials over the past 6 months prior to screening
* Active infection requiring hospitalization or treatment with parenteral antimicrobials within the 60 days prior to randomization or oral antimicrobials within the 21 days prior to enrollment
* Patient is taking >40 mg of prednisone QD
* Prior use of rituximab (or other B cell depleting agents) within 6 months of enrollment. Prior use of any B cell depleting agent greater than 6 months from enrollment is allowed if the CD19+ B cell count is within the normal reference range during screening
* Use of any investigational agent within 5 half-lives of the agent (or 6 months if the half-life is unknown) prior to enrollment
* Immunosuppressive agent use within the three months prior to enrollment
* Has received live vaccines within 2 months of enrollment
* Patient is pregnant or breast feeding, or planning to become pregnant while enrolled in the study, up to end-of-study visit
* Unable or unwilling to partake in the follow-up assessments or required protocol procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Stone, M.D., M.P.H., Principal Investigator — Rheumatology Clinic
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perugino CA, Wallace ZS, Zack DJ, Quinn SM, Poma A, Fernandes AD, Foster P, DeMattos S, Burington B, Liu H, Allard-Chamard H, Smith N, Kai X, Xing K, Pillai S, Stone JH. Evaluation of the safety, efficacy, and mechanism of action of obexelimab for the treatment of patients with IgG4-related disease: an open-label, single-arm, single centre, phase 2 pilot trial. Lancet Rheumatol. 2023 Aug;5(8):e442-e450. doi: 10.1016/S2665-9913(23)00157-1. Epub 2023 Jul 24. PMID 38251576

RESULTS

PARTICIPANT FLOW:
Groups:
- XmAb5871 5 mg/kg: 5 mg/kg weight-based dosing group
- XmAb5871 Fixed Dose: 90 mg or 180 mg fixed dose group
Period: Overall Study
Arm/Group | XmAb5871 5 mg/kg | XmAb5871 Fixed Dose
Started | 15 | 5
Completed | 12 | 4
Not Completed | 3 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XmAb5871 5 mg/kg | XmAb5871 Fixed Dose | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.57) | 51.2 (14.11) | 57.9 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 10 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 5 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 12 | 3 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 5 | 20
Serum IgG4 level at Baseline [Mean (Standard Deviation); unit: mg/dL] | 440.33 (622.990) | 858.60 (351.608) | 544.90 (588.674)
Involved Areas at Baseline [Count of Participants; unit: Participants]
  Bile Ducts | 2 | 0 | 2
  Constitutional Symptoms | 6 | 1 | 7
  Heart / Pericardium | 3 | 0 | 3
  Kidney | 5 | 1 | 6
  Lacrimal Glands | 7 | 3 | 10
  Lungs | 4 | 2 | 6
  Lymph Nodes | 10 | 4 | 14
  Nasal Cavity Lesion | 3 | 0 | 3
  Orbital Lesion | 2 | 1 | 3
  Other | 4 | 4 | 8
  Other ENT Lesions, e.g. tonsillitis, pharyngitis | 2 | 0 | 2
  Other Salivary Glands | 1 | 0 | 1
  Pancreas | 1 | 3 | 4
  Parotid Glands | 8 | 2 | 10
  Retroperitoneal Fibrosis | 1 | 1 | 2
  Sinusitis | 2 | 2 | 4
  Skin | 0 | 1 | 1
  Submandibular Glands | 9 | 3 | 12
Baseline IgG4-RD Responder Index Total Activity Score [Mean (Standard Deviation); unit: Total Activity Score] — The IgG4-RD Responder Index Total Activity Score ranges from 0 to a maximum of 162. Higher scores represent greater (i.e. worse) disease activity. A score of 0 represents no disease activity other than residual fibrosis.
  Total Activity Score | 11.5 (6.65) | 12.8 (6.42) | 11.8 (6.45)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With an Improvement in IgG4-RD Activity
Description: Improvement of disease activity as defined by a decrease of IgG4-RD responder index >= 2 points from Day 1 pre-dose disease activity score. The IgG4-RD Responder Index Total Activity Score ranges from 0 to a maximum of 162. Higher scores represent greater (i.e. worse) disease activity. A score of 0 represents no disease activity other than residual fibrosis.
Time Frame: Baseline Day 1 to Day 169
Population: Intent to Treat (ITT) Population: All patients who have received at least a partial dose of XmAb5871.
Measure: Count of Participants; unit: Participants
Arm/Group | XmAb5871 5 mg/kg | XmAb5871 Fixed Dose
Number analyzed (Participants) | 15 | 5
Participants
  Responder at Day 169 visit | 12 | 4
  Non-Responder at Day 169 visit | 2 | 0
  Not Assessed at Day 169 visit | 1 | 1

2. Secondary Outcome: Number of Patients Experiencing a Treatment-emergent Adverse Event as Assessed by CTCAE v4.3
Description: The number of patients experiencing a treatment-emergent adverse event as assessed by CTCAE v4.3 will be tabulated according to MedDRA system-organ class and preferred term, intensity and causality.
Time Frame: Baseline Day 1 to Day 197
Population: Safety Population: All patients who receive at least a partial dose of XmAb5871.
Measure: Count of Participants; unit: Participants
Arm/Group | XmAb5871 5 mg/kg | XmAb5871 Fixed Dose
Number analyzed (Participants) | 15 | 5
Participants | 13 | 5

ADVERSE EVENTS:
Time Frame: Day 1 (First Dose) through Day 197
Description: Note that due to the small total of 20 participants, the frequency threshold for reporting other adverse events applies to the total participants rather than the two defined dosing groups. Specifically, the threshold is adverse events occurring in 2 or more of 20 total participants (i.e. > 5% of 20).
Arm/Group | XmAb5871 5 mg/kg | XmAb5871 Fixed Dose
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/5
Other Adverse Events (participants affected / at risk) | 7/15 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XmAb5871 5 mg/kg (N=15) | XmAb5871 Fixed Dose (N=5)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XmAb5871 5 mg/kg (N=15) | XmAb5871 Fixed Dose (N=5)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The fixed-dose group was added by amendment to collect information on fixed IV doses with bioequivalence to subcutaneous doses planned for future studies. This group is not intended for efficacy or safety comparisons to the initial 15 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT02725476/SAP_000.pdf
  • Study Protocol (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT02725476/Prot_001.pdf